CLINICAL TRIAL: NCT06095713
Title: German Observational Multicenter Study of Patients With Fabry Disease Under Enzyme Replacement Therapy With Pegunigalsidase-alfa
Acronym: GoPEG
Status: Recruiting | Type: Observational
Sponsor: Universität Münster (Other)
Collaborators: Chiesi GmbH (Unknown)
Responsible Party: Sponsor
Other Study IDs: 11_0020WWU
Record Dates: First submitted 2023-10-10; First posted 2023-10-23 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Fabry Disease
Keywords: Pegunigalsidase-alfa
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Standard of Care: Patient treated with Pegunigalsidase-alfa according to standard of care
  Interventions: Drug: Pegunigalsidase-alfa

INTERVENTIONS:
Drug: Pegunigalsidase-alfa — Standard of care

SUMMARY:
Pegunigalsidase-alfa may represent an advance in ERT for FD, based on its unique pharmacokinetics and apparent low immunogenicity. The objective of the study is to document long term data on treatment with pegunigalsidase-alfa under "real world" conditions. 60 patients with FD (therapy-naïve or pretreated with agalsidase-alfa or agalsidase-beta) will be recruited in 8 German Fabry centers. The treatment duration/patient will be 2 years. All patients will be followed-up by the above listed Fabry expert centers.

DETAILED DESCRIPTION:
Pegunigalsidase-alfa, a novel PEGylated, covalently crosslinked form of α-galactosidase A developed as enzyme replacement therapy (ERT) for Fabry disease (FD), was designed to increase plasma half-life and reduce immunogenicity, thereby enhancing efficacy compared with available products.

The rationale of the current project is that disease progression of patients with FD can be stabilized comparable to patients under current ERT, leading to a validation of the clinical phase 3-studies and a transfer of these previous outcomes to a nationwide "real world" designed study in Germany.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, ≥18 years, diagnosed with Fabry disease.
* ERT naïve (patients with signs of organ involvement (kidney, heart and/or CNS signs) to be considered for ERT following the European Consensus Guidelines on ERT (Biegstraaten et al. 2015) or patients with neuropathic pain not controlled with pain medication or patients with GI symptoms not relieved with standard medication or ERT switch patients (under ERT for ≥12 months).
* Subjects taking ACE inhibitors, ARBs, or renin inhibitors on a stable dose for at least 4 weeks before screening.
* Subjects taking analgesics/antidepressants on a stable dose for at least 4 weeks before screening.
* Female patients must have a negative pregnancy test and use a medically accepted form of contraception throughout the study.

Exclusion Criteria:

* Patient is unwilling to give informed consent.
* Patient is unable to comply with the clinical protocol.
* Patients on dialysis.
* Patient has a clinically significant organ disease (e.g., cancer in the past 5 years) that in the opinion of the investigator would preclude participation in the trial.
* Patients with a history of organ transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with Fabry Disease
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
eGFR | yearly
  eGFR: Change in annualized eGFR slope compared with annualized eGFR slope before treatment start or switch.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Brand, MD, PhD, Principal Investigator — Universitätsklinikum Münster
Locations (8):
- Germany (8):
  - Fabry disease center Berlin - Charité - Universitätsmedizin Berlin, Berlin
  - Fabry disease center Cologne, Universitätsklinikum Köln, Cologne
  - Fabry disease center Hamburg, Universitätsklinikum Hamburg, Hamburg
  - Fabry disease center Hannover, Universitätsklinikum Hannover, Hanover
  - Fabry disease center Mainz, Universitätsmedizin Mainz, Mainz
  - Fachinternistische Gemeinschaftspraxis, Müllheim, Müllheim
  - Fabry disease center Münster, Universitätsklinikum Münster, Münster
  - Fabry disease center Würzburg, Universitätsklinikum Würzburg, Würzburg